CLINICAL TRIAL: NCT06330649
Title: The Acute Effect of and Energy Drink vs. Water Consumption on MAP, HR, and Energy Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Arlington (Other)
Responsible Party: Principal Investigator, Matthew Brothers, Professor, The University of Texas at Arlington
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2024-0095
Record Dates: First submitted 2024-03-12; First posted 2024-03-26 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Cardiovascular Diseases; Hypertension; Diet
Keywords: Energy metabolism; Arterial blood pressure; heart rate
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension | interventions — Energy Drinks

STUDY DESIGN:
Intervention Model Description: Individuals will be randomly assigned to either an experimental or a control condition.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Energy Drink (Experimental): A commercially available caffeine drink containing 200 mgs of caffeine.
  Interventions: Dietary Supplement: Energy Drink
- Water (Placebo Comparator): This will be 12 fl oz of commercially available water .
  Interventions: Other: Water Control

INTERVENTIONS:
Dietary Supplement: Energy Drink — This is a commercially available energy drink
  Arms: Energy Drink
Other: Water Control — This is a commercially available bottled water
  Arms: Water

SUMMARY:
The objective of this protocol is to investigate the effect of consumption of a commercially available energy drink beverage on blood pressure, heart rate, and energy metabolism

DETAILED DESCRIPTION:
Energy drink consumption has gained a lot in popularity and represents one of the most rapidly growing segments of the beverage industry. While regularly discussed in media outlets etc. the cardiovascular effects are not well described or well known. For example, the impacts on various cardiovascular parameters range from improved, decreased, to not impacted at all depending on the source. This can be due to a number of reasons including, study protocol design, study population tested, energy drink product used, volume consumed, etc. Accordingly, this study aims to investigate the impact of acute consumption of a standard commercially available can of energy drink beverage on the following parameters.

* Arterial blood pressure
* Heart rate
* Energy metabolism (oxygen consumption and carbon dioxide production

It is hypothesized that consumption of a 12 oz energy drink will result in modest elevations in arterial blood pressure, heart rate, and energy metabolism relative to when consuming of an equal volume of water.

ELIGIBILITY:
Inclusion Criteria:

* Between ages 18-30
* Must be free of reported cardiovascular, respiratory, and metabolic diseases.
* Must be caffeine naïve
* Must be fasted

Exclusion Criteria:

* Food allergies
* pregnant women
* Breast feeding women
* Individuals with cardiac, cardiovascular, respiratory, metabolic, and/or neurological disorders
* taking any prescription vasoactive medications
* allergies to spandex/lycra

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Peripheral blood pressure in millimeters of mercury | baseline & 30, 60, 90, 120 min following beverage consumption
  blood pressure will be measured on the upper arm using standard procedures that are done in a doctors office.
Oxygen consumption milliliters per kilogram of body weight per minute | baseline & 30, 60, 90, 120 min following beverage consumption
  This will be assessed using a metabolic cart to measure the amount of oxygen that is consumed by the body.
Heart rate in beats per minute | baseline & 30, 60, 90, 120 min following beverage consumption
  Heart will be measured using an electrocardiogram procedures that are done in a doctors office.

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Brothers, PhD, Principal Investigator — University of Texas at Arlington
Locations (1):
- UT Arlington - Science and Engineering Innovation and Research Building, Arlington, Texas, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to share IPD.